CLINICAL TRIAL: NCT05532397
Title: Evaluation of ex Vivo Drug Combination Optimization Platform in Recurrent High Grade Astrocytic Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QP/25/05/21
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Glioma, Astrocytic
Keywords: QPOP; patient-derived organoids (PDOs); TMZ/RT resistance
MeSH Terms: conditions — Astrocytoma

STUDY DESIGN:
Intervention Model Description: This is an interventional, non-randomized, open-label study. Enrolled subjects will receive QPOP-guided chemotherapy at the time of first high grade astrocytic glioma recurrence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- QPOP-guided chemotherapy (Experimental): Subjects enrolled in the study will be administered combination of chemotherapy derived from QPOP analysis based on in vitro drug screening panels which comprises anti-cancer agents which have previously been evaluated in recurrent high grade astrocytic glioma.
  Interventions: Drug: QPOP category 1; Drug: QPOP category 2

INTERVENTIONS:
Drug: QPOP category 1 — combination regimens with published data in the setting of gliomas
Drug: QPOP category 2 — combination regimens where there is published data on intracranial activity and anti-glioma effect of the individual agents either as monotherapy or in combination with other agents, and where there is published safety data on the combination

SUMMARY:
This is an interventional, non-randomized, single site study. Brain tumor samples will be collected from patients for organoids generation and subject to panel drugs screening and QPOP analysis to derive the optimal drug combinations for treatment at the time of first high grade astrocytic glioma recurrence. The investigators hypothesize that patient-derived organoids (PDOs) mimic the biological characteristics of high grade astrocytic gliomas and serve as an ideal platform for the evaluation of drug sensitivities, accurately reflecting the patient's therapeutic response to the drugs.

DETAILED DESCRIPTION:
This study aims to test the feasibility of Quadratic Phenotypic Optimization Platform (QPOP) application in high grade astrocytic glioma, by first establishing clinically relevant high grade astrocytic glioma organoid models, followed by the utility of QPOP-derived drug combinations in high grade astrocytic glioma.

The primary purpose of this study is not hypothesis testing, but to assess the feasibility of QPOP-guided therapy for recurrent high grade astrocytic glioma to be used in a larger scale study. Therefore, this study does not have a formal sample size, but rather, a set benchmarks to determine feasibility.

Specific Aim 1: To establish primary and corresponding temozolomide/radiotherapy (TMZ/RT)-resistant high grade astrocytic glioma patient-derived organoids.

Specific Aim 2: To determine the utility of QPOP (Quadratic Phenotypic Optimization Platform)-derived drug combinations in treating recurrent high grade astrocytic glioma.

Specific Aim 3: To evaluate the use of non-invasive imaging tools (Ga68-NEB PET/MRI and DCE-MRI) to track BBB permeability over time in high grade astrocytic glioma patients, and correlate this with pathological biomarkers, therapeutic response determined by follow up standard MRI and clinical outcomes.

Male and female subjects aged 21 years and above with suspected high grade astrocytic glioma planned for surgery/ biopsy followed by adjuvant chemoradiotherapy will be invited to participate in the pre-screening study. Subjects will only be enrolled in the main study if they had pathologically confirmed high grade astrocytic glioma, and received adjuvant treatment comprising standard-of-care therapy with surgery/biopsy followed by temozolomide and radiotherapy.

Pre-screening phase:

In pre-screening phase, patients will be approached for pre-screening consent at the time of first suspected diagnosis of a high grade astrocytic glioma and tumor will be harvested at the time of initial surgery/ biopsy for the generation of PDOs. Once the histological diagnosis of high grade astrocytic glioma is confirmed and the patient is planned for adjuvant temozolomide and radiotherapy, they will undergo baseline standard MRI plus Ga68-NEB PET/MRI and DCE-MRI imaging within one week of the planned radiotherapy simulation date. Patients will then undergo standard-of-care treatment for high grade astrocytic glioma with adjuvant concurrent temozolomide and radiotherapy (TMZ/RT)1, and will be evaluated by the primary oncologist routinely with clinical examination, laboratory tests and regular neuro-imaging. High grade astrocytic glioma organoids will be generated from resected tumour samples and QPOP analyses will be performed to identify specific drug combinations to guide clinical management at the time of first relapse.

Main study:

At the time of documented tumor recurrence, eligible patients will be reassessed for suitability to participate in the main study and approached for their informed consent to enter this phase of the study. During the main study, patients will receive QPOP-guided systemic therapy for the treatment of their relapsed high grade glioma and will be assessed regularly for safety and efficacy of this therapy. In addition, patients will undergo standard MRI plus investigational Ga68-NEB PET/MRI and DCE-MRI imaging prior to and 8 weeks (+/- 1 week) after QPOP-guided systemic therapy. Subsequent to this, radiological assessment of their disease will revert to standard clinical protocols with routine standard MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening:

1. Patients 21 years of age or older, with ECOG performance status 0 to 2, and with a life expectancy of more than 3 months with suspected high grade astrocytic glioma, fit for treatment comprising standard-of-care therapy with adjuvant temozolomide and radiotherapy if the diagnosis of high grade astrocytoma is pathologically confirmed.
2. Signed informed consent obtained before any study specific procedure. Subjects must be able to understand and be willing to sign the written informed consent.

   * Patients will be enrolled at the time of initial surgery but study imaging and further PDO generation will not take place if the patient is subsequently found not to meet the histological criteria or will not be receiving standard adjuvant temozolomide/ radiotherapy.

All subsequent criteria apply to the main study only:

1. Patients 21 years of age or older, with ECOG performance status 0 to 2, and life expectancy of more than 3 months with pathologically confirmed high grade astrocytic glioma, having undergone first-line standard-of-care therapy with surgery/biopsy followed by temozolomide and radiotherapy. Subjects with truncated adjuvant chemoradiotherapy may be enrolled at the Principal Investigator's discretion.
2. Documented tumor progression based on standard clinical, radiological or histological criteria, and deemed suitable for second line systemic therapy.
3. Sufficient tumor tissue available for PDO generation at baseline and at least one available or pending QPOP result.
4. Adequate organ function as defined by:

1. Bone marrow function i. Haemoglobin ≥ 9g/dl ii. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L iii. Platelet count ≥ 100 x 109/L. 2. Liver function i. Bilirubin < 2.5x upper limit of normal (ULN) ii. Alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5x ULN or < 5x ULN if liver metastases are present iii. Prothrombin time (PT) within the normal range for the institution. 3. Renal function i. Plasma creatinine <1.5x institutional ULN 5) Capable of swallowing tablets. 6) Recovery from any previous drug- or procedure-related toxicity to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 Grade 0 or 1 (except alopecia), or to baseline preceding the prior treatment.

Exclusion Criteria (both pre-screening/ main study)

1. Chemotherapy, radiotherapy, surgery, immunotherapy or other therapy within 2 weeks of study entry.
2. Pregnancy or breastfeeding at the point where systemic anti-cancer therapy is initiated. Women of childbearing potential must have a negative pregnancy test at the point where systemic anti-cancer therapy is initiated. Women of childbearing potential and men, must agree to use adequate contraception (barrier method of birth control) while on anti-cancer treatment and until at least 3 months after the last study drug administration.
3. Concurrent cancer which is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumours (Ta, Tis & T1) or any cancer curatively treated less than 5 years prior to study entry.
4. Patients with leptomeningeal dissemination of disease and/or pure spinal high grade gliomas will be excluded.
5. Kidney disease which would clinically disqualify the subject from serial MRI scans with gadolinium contrast.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Six-month progression-free survival (PFS 6) | up to 6 months
  Defined as the time from the start of study treatment to documented progression of disease or death; PFS6 refers to the percentage of patients who are alive and free of high grade astrocytic glioma progression at 6 months.

SECONDARY OUTCOMES:
Radiological response at follow up MRI | Up to 6 months
  The determination of radiographic response is as per the Response Assessment in Neuro-Oncology (RANO) criteria.
Twelve-month overall survival (OS12) | Up to 12 months
  OS is defined as the length of time from the start of study treatment, that patients diagnosed with the disease are still alive. OS12 refers to the percentage of patients who are alive at 12 months.
Number of participant with treatment related haematological and non-haematological toxicities | Up to 6 months
  As defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Wong, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - Department of Hematology-Oncology, National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Brandes AA, Basso U, Reni M, Vastola F, Tosoni A, Cavallo G, Scopece L, Ferreri AJ, Panucci MG, Monfardini S, Ermani M; Gruppo Italiano Cooperativo di Neuro-Oncologia. First-line chemotherapy with cisplatin plus fractionated temozolomide in recurrent glioblastoma multiforme: a phase II study of the Gruppo Italiano Cooperativo di Neuro-Oncologia. J Clin Oncol. 2004 May 1;22(9):1598-604. doi: 10.1200/JCO.2004.11.019. PMID 15117981
- [Background] Chamberlain MC, Tsao-Wei DD. Salvage chemotherapy with cyclophosphamide for recurrent, temozolomide-refractory glioblastoma multiforme. Cancer. 2004 Mar 15;100(6):1213-20. doi: 10.1002/cncr.20072. PMID 15022289
- [Background] Chatzellis E, Angelousi A, Daskalakis K, Tsoli M, Alexandraki KI, Wachula E, Meirovitz A, Maimon O, Grozinsky-Glasberg S, Gross D, Kos-Kudla B, Koumarianou A, Kaltsas G. Activity and Safety of Standard and Prolonged Capecitabine/Temozolomide Administration in Patients with Advanced Neuroendocrine Neoplasms. Neuroendocrinology. 2019;109(4):333-345. doi: 10.1159/000500135. Epub 2019 Jun 3. PMID 31167197
- [Background] Field KM, Simes J, Nowak AK, Cher L, Wheeler H, Hovey EJ, Brown CS, Barnes EH, Sawkins K, Livingstone A, Freilich R, Phal PM, Fitt G; CABARET/COGNO investigators; Rosenthal MA. Randomized phase 2 study of carboplatin and bevacizumab in recurrent glioblastoma. Neuro Oncol. 2015 Nov;17(11):1504-13. doi: 10.1093/neuonc/nov104. Epub 2015 Jun 30. PMID 26130744
- [Background] Forsyth P, Cairncross G, Stewart D, Goodyear M, Wainman N, Eisenhauer E. Phase II trial of docetaxel in patients with recurrent malignant glioma: a study of the National Cancer Institute of Canada Clinical Trials Group. Invest New Drugs. 1996;14(2):203-6. doi: 10.1007/BF00210791. PMID 8913841
- [Background] Francesconi AB, Dupre S, Matos M, Martin D, Hughes BG, Wyld DK, Lickliter JD. Carboplatin and etoposide combined with bevacizumab for the treatment of recurrent glioblastoma multiforme. J Clin Neurosci. 2010 Aug;17(8):970-4. doi: 10.1016/j.jocn.2009.12.009. Epub 2010 Jun 11. PMID 20541421
- [Background] Friedman HS, Petros WP, Friedman AH, Schaaf LJ, Kerby T, Lawyer J, Parry M, Houghton PJ, Lovell S, Rasheed K, Cloughsey T, Stewart ES, Colvin OM, Provenzale JM, McLendon RE, Bigner DD, Cokgor I, Haglund M, Rich J, Ashley D, Malczyn J, Elfring GL, Miller LL. Irinotecan therapy in adults with recurrent or progressive malignant glioma. J Clin Oncol. 1999 May;17(5):1516-25. doi: 10.1200/JCO.1999.17.5.1516. PMID 10334539
- [Background] Lu G, Rao M, Zhu P, Liang B, El-Nazer RT, Fonkem E, Bhattacharjee MB, Zhu JJ. Triple-drug Therapy With Bevacizumab, Irinotecan, and Temozolomide Plus Tumor Treating Fields for Recurrent Glioblastoma: A Retrospective Study. Front Neurol. 2019 Jan 31;10:42. doi: 10.3389/fneur.2019.00042. eCollection 2019. PMID 30766509
- [Background] Wick W, Gorlia T, Bendszus M, Taphoorn M, Sahm F, Harting I, Brandes AA, Taal W, Domont J, Idbaih A, Campone M, Clement PM, Stupp R, Fabbro M, Le Rhun E, Dubois F, Weller M, von Deimling A, Golfinopoulos V, Bromberg JC, Platten M, Klein M, van den Bent MJ. Lomustine and Bevacizumab in Progressive Glioblastoma. N Engl J Med. 2017 Nov 16;377(20):1954-1963. doi: 10.1056/NEJMoa1707358. PMID 29141164
- [Background] Grisanti S, Ferrari VD, Buglione M, Agazzi GM, Liserre R, Poliani L, Buttolo L, Gipponi S, Pedersini R, Consoli F, Panciani P, Roca E, Spena G, Triggiani L, Berruti A; Gruppo Neuro-Oncologico Bresciano. Second line treatment of recurrent glioblastoma with sunitinib: results of a phase II study and systematic review of literature. J Neurosurg Sci. 2019 Aug;63(4):458-467. doi: 10.23736/S0390-5616.16.03874-1. Epub 2016 Sep 28. PMID 27680966
- [Background] Kreisl TN, Lassman AB, Mischel PS, Rosen N, Scher HI, Teruya-Feldstein J, Shaffer D, Lis E, Abrey LE. A pilot study of everolimus and gefitinib in the treatment of recurrent glioblastoma (GBM). J Neurooncol. 2009 Mar;92(1):99-105. doi: 10.1007/s11060-008-9741-z. Epub 2008 Nov 19. PMID 19018475
- [Background] Lassman AB, Wen PY, van den Bent MJ, Plotkin SR, Walenkamp AME, Green AL, Li K, Walker CJ, Chang H, Tamir S, Henegar L, Shen Y, Alvarez MJ, Califano A, Landesman Y, Kauffman MG, Shacham S, Mau-Sorensen M. A Phase II Study of the Efficacy and Safety of Oral Selinexor in Recurrent Glioblastoma. Clin Cancer Res. 2022 Feb 1;28(3):452-460. doi: 10.1158/1078-0432.CCR-21-2225. Epub 2021 Nov 2. PMID 34728525
- [Background] Lesueur P, Lequesne J, Grellard JM, Dugue A, Coquan E, Brachet PE, Geffrelot J, Kao W, Emery E, Berro DH, Castera L, Goardon N, Lacroix J, Lange M, Capel A, Leconte A, Andre B, Leger A, Lelaidier A, Clarisse B, Stefan D. Phase I/IIa study of concomitant radiotherapy with olaparib and temozolomide in unresectable or partially resectable glioblastoma: OLA-TMZ-RTE-01 trial protocol. BMC Cancer. 2019 Mar 4;19(1):198. doi: 10.1186/s12885-019-5413-y. PMID 30832617
- [Derived] Toh TB, Thng DKH, Bolem N, Vellayappan BA, Tan BWQ, Shen Y, Soon SY, Ang YLE, Dinesh N, Teo K, Nga VDW, Low SW, Khong PL, Chow EK, Ho D, Yeo TT, Wong ALA. Evaluation of ex vivo drug combination optimization platform in recurrent high grade astrocytic glioma: An interventional, non-randomized, open-label trial protocol. PLoS One. 2024 Jul 26;19(7):e0307818. doi: 10.1371/journal.pone.0307818. eCollection 2024. PMID 39058662